CLINICAL TRIAL: NCT03905837
Title: Impact of the Administration of Intravenous or Paravertebral Lidocaine in Continuous Perfusion During the Intraoperative Period of Lung Resection Surgery on the Appearance of Postoperative Complications
Brief Title: Impact of Lidocaine Administration on Postoperative Complications During Lung Resection Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Francisco Andres de la Gala (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Francisco Andres de la Gala, Anesthesiologist. MD. PhD, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IGMFGG-2016
Record Dates: First submitted 2019-03-26; First posted 2019-04-05 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Lung Diseases; Lung Inflammation; Lung Injury, Acute; Postoperative Complications
Keywords: lidocaine; postoperative complications; thoracic surgery
MeSH Terms: conditions — Lung Diseases; Pneumonia; Acute Lung Injury; Postoperative Complications | interventions — Lidocaine; Remifentanil

STUDY DESIGN:
Intervention Model Description: Unicentric, randomized, blind and controlled phase IV Clinical trial of three parallel groups.
  Randomization: Patients will be randomized into three groups (ratio 1: 1: 1): intravenous lidocaine and paravertebral saline (group 1), intravenous and paravertebral saline solution with lidocaine (group 2) and intravenous remifentanil and paravertebral saline solution (group 3) ). The randomization will be carried out through the EPIDAT 3.1 program prior to the recruitment of the first patient and the randomization codes will be kept in a sealed envelope with the number on the outside of the envelope. Patients will be followed from the day of hospital admission until hospital discharge and after 30 days of surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be carried out through the EPIDAT 3.1 program. Randomization codes will be obtained prior to the recruitment of the first patient and will be kept in a sealed envelope with numbering on the outside of the envelope. The operating room anesthesiologist will receive the assigned medication from the corresponding group with the only identification of intravenous perfusion and paravertebral perfusion, without having knowledge of the group to which the patient belongs.
  Bias control: The anesthesiologist responsible for the intraoperative management of the patient, the physician responsible for postoperative control in the postoperative care unit and the guard physician who will perform the cognitive dysfunction test preoperative and postoperative and the follow up until the month of surgery will be blind to the technique used, as well as those responsible for the analysis of the biological samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine IV (Experimental): Group 1: intravenous lidocaine and paravertebral saline (SF). In this group during intraoperative anesthetic maintenance, a continuous intravenous infusion of lidocaine at 1.5mg/kg/h until the end of surgery and perfusion of 0.9% SF through the intraoperative paravertebral catheter at a rate of 0.1ml/kg/h will be administered.
  Interventions: Drug: Lidocaine
- Lidocaine PV (Experimental): Group 2: intravenous SF and paravertebral lidocaine. During anesthesia maintenance, a continuous intravenous infusion of 0.9% SF and an infusion of 2% lidocaine will be administered through the intraoperative paravertebral catheter at a rate of 0.1 ml/kg/h.
  Interventions: Drug: Lidocaine
- no lidocaine (Active Comparator): Group 3: intravenous remifentanil and paravertebral SF. During the maintenance of anesthesia, a continuous intravenous infusion of remifentanil at a rate of 0.1 mg/kg/min until the end of surgery and an infusion of 0.9% SF through the intraoperative paravertebral catheter at a rate of 0.1 ml / kg / h.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Lidocaine — Intravenous or paravertebral lidocaine
  Other Names: Lignocaine; N-(2,6-dimethylphenyl)-N2,N2-diethylglycinamide
  Arms: Lidocaine IV; Lidocaine PV
Drug: Remifentanil — intravenous remifentanil
  Other Names: methyl 1-(2-methoxycarbonylethyl)-4-(phenyl-propanoyl-amino)-piperidine-4-carboxylate
  Arms: no lidocaine

SUMMARY:
The purpose of this study is to analyze the impact of the intravenous (IV) or paravertebral (PV) lidocaine administration during the intraoperative period of lung resection surgery on the appearance of postoperative complications. We design a randomized, controlled and blinded study to be performed in 153 patients with 3 arms: 1) Lidocaine IV + PV saline 2) saline IV + PV lidocaine, 3) remifentanil IV + PV saline. Perioperative analysis of inflammatory biomarkers in bronchoalveolar lavage and serum. Follow-up of the postoperative course, especially the appearance of postoperative complications according to the revised Clavien-Dindo classification for thoracic surgery, as well as other relevant clinical results.

DETAILED DESCRIPTION:
Postoperative pulmonary complications continue to be one of the main causes of morbidity, mortality and increase in hospital stay in patients undergoing surgical procedures requiring anesthesia. Its incidence in lung resection surgery is greater than in other non-cardiac major surgeries due to damage of structures related to respiratory function.

Furthermore, during lung resection surgery there is an exaggerated pulmonary inflammatory response related to the use of one-lung ventilation and / or the lung damage produced by the collapse of the operated lung as well as the surgical manipulation itself.

Recently, in a clinical trial on 180 patients (NCT 02168751), our researcher group observed that the attenuation of the pulmonary inflammatory response through the use of halogenated anesthetic agents, was related to a decrease in the appearance of postoperative pulmonary complications after lung resection surgery. In addition, the presence, in bronchoalveolar lavages, of elevated levels of tumor necrosis factor-alpha, interleukine(IL)-6 and the IL-6 / IL10 ratio were independent predictors of the risk of developing postoperative pulmonary complications.

Lidocaine is a local anesthetic that blocks nerve conduction by blocking sodium channels. In addition it has been known for experimental and clinical studies of its immunomodulatory properties.

Clinical studies performed in different surgeries show that a continuous intravenous infusion of lidocaine during surgery is associated with a lower inflammatory response assessed by monitoring plasma cytokines, as well as less postoperative pain, a shorter duration of postoperative paralytic ileus and a early hospital discharge.

Currently, there is no clinical study that has evaluated the role of intravenous lidocaine on the pulmonary inflammatory response and the subsequent lung damage that inevitably occurs during lung resection surgery with periods of one lung ventilation.

Currently, some experts are proposing the replacement of thoracic epidural and paravertebral analgesia by the intravenous infusion of lidocaine and minor analgesics, for fast-track programs, based on their analgesic and anti-inflammatory capacity and on avoiding the risks inherent in the insertion of an epidural or paravertebral catheter.

Hypothesis: The administration of intravenous or paravertebral lidocaine during lung resection surgery attenuates the exaggerated inflammatory response that inevitably occurs in this surgical intervention. The lower expression of pro-inflammatory mediators will be associated with a lower rate of postoperative complications that are related to the perioperative inflammatory process.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes undergoing lung resection surgery at the Thoracic Surgery Service at the Gregorio Maranón hospital.
* Patients who voluntarily accept to participate in the study and sign the informed consent
* Age> 18 years and legally capable
* Scheduled surgery.
* Functional respiratory tests with forced expiratory volume at one second > 50% or forced vital capacity > 50% preoperatively performed on these patients routinely.
* Not having been on chronic treatment with oral corticosteroids or immunosuppressants three months before surgery.
* Patients without previous history of liver disease.

Exclusion Criteria:

* Pregnancy and lactation
* Known hypersensitivity to amide-type local anesthetics.
* Transfusion of blood products in the previous 10 days.
* Impossibility of performing mechanical ventilation for pulmonary protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | up to 30 days after intervention
  to compare the proportion of patients included in the different scales of the Clavien-Dindo classification of postoperative complications reviewed for thoracic surgery in the three groups of patients. Patients will be followed from the day of hospital admission until hospital discharge and up to 30 days after the surgery

SECONDARY OUTCOMES:
gas exchange | 24 hours
  Compare the gas exchange (PaO2 / FiO2) at 24 hours after the intervention between the three groups of the study.
Differences between three groups in Inflammatory biomarkers (IL 1, IL 2, IL 6, IL 8, IL 10, TNF alpha, MCP-1) measure in serum and bronchoalveolar lavage during 24 hours after the surgery. | up to 24 hours of intervention
  To evaluate the effect of intravenous lidocaine on the inflammatory response in lung resection surgery by measuring the inflammatory biomarkers (Interleukin(IL) 1, IL 2, IL 6, IL8, IL 10, tumor necrosis factor alfa and monocyte chemoattractant protein) in serum and in bronchoalveolar lavage, compared to the other two groups of patients. Blood samples are taken at the beginning of the surgery, at the end of the one lung ventilation, and at 24 hours postoperatively. Bronchoalveolar lavage is done just before the beginning of one lung ventilation and at the end of one lung ventilation
Analgesic requirements of opioids in the first 24 hours after the surgery | 24 hours
  To compare the analgesic requirements of opioids in the immediate postoperative period (first 24 hours after the surgery) between the three groups of the study. When patients will be admitted in the postoperative care Unit a patient controlled analgesia pump of intravenous morphine 0,1% (bolus of 1mg) will be connected. The total dose of morphine self-administered by the patient in the first 24 hours after surgery will be recorded.
Special Care Units stay | up to 30 days after intervention
  To compare the average stay (measure in hours) in Special Care Units among the three groups of the study
Hospital stay | up to 30 days after intervention
  To compare the average hospital stay (measure in days) among the three groups of the study
Re-admissions in Special Care Units | up to 30 days after intervention
  To compare the number of re-admissions in Special Care Units among the three groups of the study in the 30 days after the intervention.
Postoperative cognitive dysfunction measure by mini mental state examination | up to 3 days after intervention
  To analyze the incidence of postoperative cognitive dysfunction (POCD) in the three groups by comparing the mini mental state examination performed at admission and 3 days after the intervention.
Neuro-inflammatory response measure by the synthesis of protein S-100 beta in serum | up to 24 hours after intervention
  To evaluated the neuro-inflammatory response by the synthesis of protein S-100 beta measured in serum in the first 24 hours postoperatively in the three groups of patients. Blood samples are taken at the beginning of the surgery, at the end of the one lung ventilation, and at 24 hours postoperatively
Neuro-inflammatory response measure by the synthesis of neuronal specific enolase in serum | up to 24 hours after intervention
  To evaluated the neuro-inflammatory response by the synthesis of neuronal specific enolase measured in serum in the first 24 hours postoperatively in the three groups of patients. Blood samples are taken at the beginning of the surgery, at the end of the one lung ventilation, and at 24 hours postoperatively
Neuro-inflammatory response measure by the synthesis of glial fibrillary acidic protein | up to 24 hours after intervention
  To evaluated the neuro-inflammatory response by the synthesis of glial fibrillary acidic protein measured in serum in the first 24 hours postoperatively in the three groups of patients. Blood samples are taken at the beginning of the surgery, at the end of the one lung ventilation, and at 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Francisco de la Gala, MD PhD, Principal Investigator — Hospital Gregorio Maranon
Locations (1):
- Hospital Gregorio Maranon, Madrid, Spain

REFERENCES:
- [Derived] de la Gala F, de la Fuente E, Pineiro P, Reyes A, Duque P, Sanchez-Pedrosa G, Martinez-Gascuena D, Vara E, Rancan L, Simon C, Hortal J, Garutti I. Effect of intraoperative paravertebral or intravenous lidocaine infusion on postoperative complications and inflammation after lung resection surgery: a randomised controlled trial. Br J Anaesth. 2025 Nov;135(5):1297-1306. doi: 10.1016/j.bja.2025.05.059. Epub 2025 Sep 1. PMID 40897588
- [Derived] De la Gala F, Pineiro P, Reyes A, Simon C, Vara E, Rancan L, Huerta LJ, Gonzalez G, Benito C, Munoz M, Grande P, Paredes SD, Aznar PT, Perez A, Martinez D, Higuero F, Sanz D, De Miguel JP, Cruz P, Olmedilla L, Lopez Gil E, Duque P, Sanchez-Pedrosa G, Valle M, Garutti I. Effect of intraoperative paravertebral or intravenous lidocaine versus control during lung resection surgery on postoperative complications: A randomized controlled trial. Trials. 2019 Nov 6;20(1):622. doi: 10.1186/s13063-019-3677-9. PMID 31694684